CLINICAL TRIAL: NCT02248103
Title: Comparison of Autogenous Periosteal Pedicle Graft and Collagen Membrane in Management of Periodontal Intrabony Defects: A Randomized Controlled Clinical Trial.
Brief Title: Comparison of Autogenous Periosteal Pedicle Graft and Collagen Membrane in Management of Periodontal Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of periodontology, faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPP graft_GTR
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- periosteal pedicle graft (Experimental): autogenous marginal periosteal pedicle graft harvested by partial thickness periodontal flap.
  Interventions: Procedure: Periosteal pedicle graft
- Bioresorbable collagen membrane (Active Comparator): Equine Achilles tendon collagen barrier membrane
  Interventions: Biological: Bioresorbable collagen membrane

INTERVENTIONS:
Procedure: Periosteal pedicle graft — Autogenous pedicle graft harvested from the periosteum
  Arms: periosteal pedicle graft
Biological: Bioresorbable collagen membrane — Biocollagen is a thin equine Achilles tendon collagen barrier membrane used for guided tissue regeneration
  Arms: Bioresorbable collagen membrane

SUMMARY:
A clinical and radiographic evaluation of autogenous periosteal pedicle graft in comparison with collagen membrane for management of periodontal intrabony defects.

DETAILED DESCRIPTION:
Twenty patients suffering from advanced chronic periodontitis were included in this randomized controlled clinical trial. Each subject contributed matched pairs of two- or three-walled intrabony defects. Each pair of periodontal defects were randomly assigned into the experimental group; periosteal pedicle graft guided tissue membrane or the positive control group; bioresorbable collagen guided tissue regeneration membrane. Clinical and radiographic parameters were recorded at baseline and at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Severe chronic periodontitis patients with at least two sites with pocket depth ≥ 6 mm and clinical attachment level ≥ 5 mm, with radiographic evidence of bone loss 2- or 3-wall intrabony defect depth ranging from 3 to 6 mm as detected in periapical radiographs
* The facial surface of teeth adjacent to the interproximal defect should be free of extensive recession and marginal bone loss, with at least a 4 to 5 mm band of keratinized gingiva to allow for periosteal manipulation

Exclusion Criteria:

* Pregnant women
* Subjects had <22 permanent teeth
* Having any given systemic disease
* Taking any type of medication and/or antibiotic therapy during the 3 months before the study
* Received periodontal treatment within the past 12 months
* Current or former smokers

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noha Ghallab, M.D., Principal Investigator — Associate Professor of periodontology faulty of oral and dental medicine Cairo Unv.

REFERENCES:
- [Result] Singhal R, Nandlal, Kumar A, Rastogi P. Role of space provision in regeneration of localized two-wall intrabony defects using periosteal pedicle graft as an autogenous guided tissue membrane. J Periodontol. 2013 Mar;84(3):316-24. doi: 10.1902/jop.2012.110734. Epub 2012 May 21. PMID 22612365
- [Result] Gamal AY, Mailhot JM. A novel marginal periosteal pedicle graft as an autogenous guided tissue membrane for the treatment of intrabony periodontal defects. J Int Acad Periodontol. 2008 Oct;10(4):106-17. PMID 19055224
- [Result] Paolantonio M, Femminella B, Coppolino E, Sammartino G, D'Arcangelo C, Perfetti G, Perinetti G. Autogenous periosteal barrier membranes and bone grafts in the treatment of periodontal intrabony defects of single-rooted teeth: a 12-month reentry randomized controlled clinical trial. J Periodontol. 2010 Nov;81(11):1587-95. doi: 10.1902/jop.2010.100094. Epub 2010 Jun 28. PMID 20583915
- [Result] Bunyaratavej P, Wang HL. Collagen membranes: a review. J Periodontol. 2001 Feb;72(2):215-29. doi: 10.1902/jop.2001.72.2.215. PMID 11288796
- [Result] Stoecklin-Wasmer C, Rutjes AW, da Costa BR, Salvi GE, Juni P, Sculean A. Absorbable collagen membranes for periodontal regeneration: a systematic review. J Dent Res. 2013 Sep;92(9):773-81. doi: 10.1177/0022034513496428. Epub 2013 Jul 10. PMID 23842107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Periosteal Pedicle Graft | Bioresorbable Collagen Membrane
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Periosteal Pedicle Graft | Bioresorbable Collagen Membrane | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.81 (8.3) | 37.81 (8.3) | 37.81 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Attachment Level
Description: Estimation of clinical attachment level in chronic periodontitis patients at baseline and 6 months after guided tissue regeneration
Time Frame: Baseline and 6 months
Population: defects
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Periosteal Pedicle Graft | Bioresorbable Collagen Membrane
Number analyzed (Participants) | 10 | 10
mm
  Baseline CAL | 6.42 (0.56) | 6.15 (0.98)
  CAL after 6 months | 3.52 (0.44) | 3.6 (0.57)

2. Secondary Outcome: Pocket Depth
Description: Estimation of pocket depth in chronic periodontitis patients at baseline and 6 months after guided tissue regeneration
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Periosteal Pedicle Graft | Bioresorbable Collagen Membrane
Number analyzed (Participants) | 10 | 10
mm
  Baseline PD | 6.92 (0.76) | 6.82 (1.1)
  PD after 6 months | 3.17 (0.65) | 3.15 (0.67)

3. Secondary Outcome: Bone Defect Area
Description: linear measurements collected from a digital radiography program to estimate percentage of defect fill.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: "mm^2"
Arm/Group | Periosteal Pedicle Graft | Bioresorbable Collagen Membrane
Number analyzed (Participants) | 10 | 10
"mm^2"
  Baseline bone defect area | 8.37 (4.13) | 9.25 (3.23)
  Bone defect area after 6 months | 4.42 (0.72) | 5.7 (2.99)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Periosteal Pedicle Graft | Bioresorbable Collagen Membrane
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No